CLINICAL TRIAL: NCT00063180
Title: Remote Effects of Stroke on Cerebral Metabolism. Evaluation With Positron Emission Tomography and Proton Magnetic Resonance Spectroscopy
Brief Title: Evaluating the Remote Effects of Stroke With MRI and PET Scans
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030224; 03-N-0224
Record Dates: First submitted 2003-06-20; First posted 2003-06-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-20

CONDITIONS: Cerebrovascular Accident
Keywords: Diaschisis; Glucose; GABA; N-Acetylaspartate; Glutamate; Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke; Diaschisis

SUMMARY:
Patients with stroke sometimes have a condition called diaschisis, a loss of function in a part of the brain located some distance from the original stroke-injury site. Doctors do not know why this happens.

The purpose of this study is to get a better understanding as to why diaschisis occurs by studying people who have experienced a stroke and people who have aged in good health.

Forty-four participants who are older than 40 year of age will be enrolled in this study-18 healthy people and 26 stroke patients. They will have 3 to 4 study visits. The first visit will involve a medical history and a physical and neurological exam. Participants will then have a magnetic resonance imaging (MRI) scan, either on the first visit or on a later day. On the next visit, they will undergo a position emission tomography (PET) scan. Finally, they will return for another MRI scan.

DETAILED DESCRIPTION:
Objective: Following a stroke, not only is there dysfunction of the lesioned area, but there is also remote functional depression of non-lesioned areas. This functional depression, called diaschisis, likely contributes to the functional deficit of the patient.

The objective of this study is to obtain a better understanding of the pathophysiology of diaschisis with the integrated methods of neuroimaging (positron emission tomography (PET) and proton magnetic resonance spectroscopy (H-MRS)).

Study population: We will recruit patients with subcortical stroke in the subacute state and in the chronic state, and normal controls.

Design: The stroke lesion will be the basal ganglia, internal capsule, thalamus, or cerebellum. The frontal cortex, including the motor cortex, is chosen as a remote area. Neurochemical changes in the diaschitic area will be investigated by measuring the glucose metabolic rate with PET, and concentrations of neurochemically important metabolites, such as gamma-aminobutyric acid (GABA) and glutamate, with H-MRS.

Outcome measures: Metabolic change in the diaschitic areas relative to the contra-lateral unaffected side will be calculated as a laterality index. First, this index will be compared among patient groups and control group. As a second analysis, the relationship of glucose metabolism measured by PET and concentrations of the metabolites detected by H-MRS will be evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will have a clinically and radiologically documented stroke in the subacute (2 weeks to 6 months to after onset) or the chronic state (more than 6 months after onset), having a lesion in subcortical regions including the basal ganglia, thalamus, internal capsule, or a combination of these structures, or cerebellum unilaterally. These lesions can extend to the surrounding areas, however not including the cerebral areas where H-MRS ROI will be located. Both ischemic infarction and hemorrhage will be included; however, in cases of hemorrhage, we will exclude cases with deformation in the cerebral hemisphere due to mass effect of the hemorrhage, hydrocephalus, or extension to the ventricles. Patients will be 18 years of age or older.

Healthy controls entering the study must be free of serious somatic disease as determined by a standard physical and neurological examination. Controls will be aged over 18 years.

Female patients and controls of child bearing potential will have a pregnancy test and specific interview prior to the study to ensure that pregnant patients will not participate in the study. Both patients and controls will be asked to abstain from alcohol for one week before each of the PET and H-MRS scans.

EXCLUSION CRITERIA:

A. Patients with MRI findings consistent with brain tumors, trauma or AVMs will be excluded.

B. Patients with multiple stroke lesions will be excluded, except for prior asymptomatic lacunar infarctions or stroke lesions which are not known to cause diaschisis in the frontal cortex (occipital cortex).

C. Patients with severe stenosis (greater than 70%) or occlusion in internal cervical arteries and in the proximal portions of middle or frontal cerebral arteries detected by angiography or MRA will be excluded. Subjects with medical disorders which can affect the concentration of cerebral metabolites, including renal failure, hepatic failure and untreated electrolyte abnormality will be excluded. Subjects with poorly controlled diabetes mellitus (casual plasma glucose concentration greater than or equal to 200 mg per dL (11.1 mmol per L) or fast plasma glucose concentration greater than or equal to 126 mg per dL (7.0 mmol per L) will be excluded. Subjects who are taking sleeping drugs or tranquilizers will be asked to stop taking them for two days prior to each of the PET and H-MRS scans.

D. Subjects with a pre-stroke history of schizophrenia or bipolar disorders will be excluded.

E. Subjects with implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may be contraindicated or prevent the acquisition of MRI.

F. Subjects with cancer will be excluded.

G. Patients not capable of giving an informed consent will be excluded

H. Ethnic origin and race will not be biased for inclusion.

Participation of children:

Children will be excluded from the study because we need to study a homogeneous group of subjects by age and developmental changes in metabolites will complicate this study. Additionally, young children will not be sufficiently cooperative for the long periods of testing. Moreover, the radiation dose of the PET studies would subject them to relatively greater risk than the adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-06-19; Study Completion 2009-04-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chang L, Cloak CC, Ernst T. Magnetic resonance spectroscopy studies of GABA in neuropsychiatric disorders. J Clin Psychiatry. 2003;64 Suppl 3:7-14. PMID 12662128
- [Background] Chu WJ, Mason GF, Pan JW, Hetherington HP, Liu HG, San Pedro EC, Mountz JM. Regional cerebral blood flow and magnetic resonance spectroscopic imaging findings in diaschisis from stroke. Stroke. 2002 May;33(5):1243-8. doi: 10.1161/01.str.0000015240.75199.be. PMID 11988598
- [Background] Brooks JC, Roberts N, Kemp GJ, Gosney MA, Lye M, Whitehouse GH. A proton magnetic resonance spectroscopy study of age-related changes in frontal lobe metabolite concentrations. Cereb Cortex. 2001 Jul;11(7):598-605. doi: 10.1093/cercor/11.7.598. PMID 11415962